CLINICAL TRIAL: NCT06226844
Title: Evaluation of the Value of Music Therapy (BeatMove Device) in a 3-month Outpatient Walking Rehabilitation Programme for Patients With Obliterative Arterial Disease of the Lower Limbs (AOMI) at the Stress Ischaemia Stage.
Brief Title: Can the BeatMove Device Help Patients With Obliterative Arterial Disease of the Lower Limbs?
Acronym: LEGS GO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ID-RCB 2023-A02245-40
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Atheromatous; Lower Limb Ischemia; Artery Disease
Keywords: Rehabilitation; Music therapy
MeSH Terms: conditions — Plaque, Atherosclerotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group : PEMA SHAM (Sham Comparator): Patients on rehabilitation using the BeatMove device in sham mode
  Interventions: Device: Sham BeatMove
- Experimental group : PEMA BeatMove (Experimental): Patients on rehabilitation using the BeatMove device
  Interventions: Device: Music therapy walking program

INTERVENTIONS:
Device: Music therapy walking program — In the experimental group (PEMA BeatMove), patients will benefit from an outpatient walking training program with app-based performance monitoring, combined with music therapy (BeatMove device). The program comprises 36 walking training sessions, with 30
  Arms: Experimental group : PEMA BeatMove
Device: Sham BeatMove — Ambulatory gait training program with performance monitoring via an app, combined with sham music therapy (BeatMove device). The program includes 36 gait training sessions, each lasting 30 minutes. Patients will complete three walking sessions per week for three months.
  Arms: Control group : PEMA SHAM

SUMMARY:
Vascular rehabilitation for arteriopathy of the lower limbs remains little known in France, despite its good results. There are very few rehabilitation centres, and they are overcrowded and expensive. Outpatient walking rehabilitation is under-used, despite recommendations (4). One of the difficulties is getting patients to adhere to the treatment sufficiently and for a long time. According to the Fédération Française de Musicothérapie (FFM), this is a care practice based on sound or musical mediation with the aim of supporting, accompanying or re-educating a patient. Music is used as a means of expression, communication, structuring and relational analysis.The benefits of music therapy for our bodies and our behavior are numerous, including improvements in cognitive functions (attention, memory), psychomotor functions (agility, mobility, coordination) and social-emotional functions (healthymind website 10/03/2021).

DETAILED DESCRIPTION:
Atheromatous obliterative arterial disease of the lower limbs at the stage of exertional ischaemia is characterised by intermittent claudication, defined as pain in the lower limbs on walking, forcing the patient to stop for a few minutes after a distance that varies according to the severity of the arterial damage. Physical exercise, and walking training in particular, plays a fundamental role in the management of patients with arterial disease. The beneficial effects of exercise are well known. A recent Cochrane review showed that exercise improves pain-free walking distance and maximum walking distance by at least 100% in patients with arterial hypertension (2). Exercise also significantly reduces total and cardiovascular mortality (3).

In the case of intermittent claudication, medical treatment with supervised vascular rehabilitation is recommended in rehabilitation centres or on an outpatient basis. Vascular rehabilitation for arteriopathy of the lower limbs remains little known in France, despite its good results. There are very few rehabilitation centres, and they are overcrowded and expensive. Outpatient walking rehabilitation is under-used, despite recommendations (4). One of the difficulties is getting patients to adhere to the treatment sufficiently and for a long time.

Musico therapy : According to the Fédération Française de Musicothérapie (FFM), this is a care practice based on sound or musical mediation with the aim of supporting, accompanying or re-educating a patient. Music is used as a means of expression, communication, structuring and relational analysis.

The benefits of music therapy for our bodies and our behavior are numerous, including improvements in cognitive functions (attention, memory), psychomotor functions (agility, mobility, coordination) and social-emotional functions (healthymind website 10/03/2021).

ELIGIBILITY:
Inclusion Criteria:

* Patient with stage II arterial obliteration of the lower limbs (Leriche and Fontaine classification) with exertional claudication
* Systolic Pressure Index at the toe < 0.7 but absolute value > 30 mmHg
* Steno-occlusive lesions on arterial Doppler ultrasound examination of the lower limbs
* Patient on an optimised vasculoprotective medical treatment (statin, antiplatelet agent, ACE inhibitor/ARB II)
* Patient who is a beneficiary or entitled beneficiary of a health insurance scheme
* Patient able to understand, write and read French
* Patient who has given free and informed consent

Exclusion Criteria:

* Patients using walking aids (cane, wheelchair)
* Amputation
* Patient with a walking perimeter < 150 m
* Hearing or visual impairment
* Chronic ischaemia
* Trophic disorders
* Orthopaedic or vascular MI surgery planned within 3 months
* Major cardiovascular co-morbidities (MI < 3 months or unstable angina)
* Pregnant, breast-feeding or parturient women
* Patients under court protection, guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Benefit of music therapy (delivered by the BeatMove device) in a three-month outpatient walking rehabilitation: Experimental group. | Week 4
  Maximum walking distance defined as the walking distance to the point of maximum muscular pain requiring stopping, during a treadmill test.
  Patients will have to do 3 walking sessions per week for a total duration of 12 weeks.
Benefit of music therapy (delivered by the BeatMove device) in a three-month outpatient walking rehabilitation: Sham group. | Week 4
  Maximum walking distance defined as the walking distance to the point of maximum muscular pain requiring stopping, during a treadmill test.
  Patients will have to do 3 walking sessions per week for a total duration of 12 weeks.
Benefit of music therapy (delivered by the BeatMove device) in a three-month outpatient walking rehabilitation: Experimental group. | Week 8
  Maximum walking distance defined as the walking distance to the point of maximum muscular pain requiring stopping, during a treadmill test.
  Patients will have to do 3 walking sessions per week for a total duration of 12 weeks.
Benefit of music therapy (delivered by the BeatMove device) in a three-month outpatient walking rehabilitation: Sham group. | Week 8
  Maximum walking distance defined as the walking distance to the point of maximum muscular pain requiring stopping, during a treadmill test.
  Patients will have to do 3 walking sessions per week for a total duration of 12 weeks.
Benefit of music therapy (delivered by the BeatMove device) in a three-month outpatient walking rehabilitation: Experimental group. | Week 12
  Maximum walking distance defined as the walking distance to the point of maximum muscular pain requiring stopping, during a treadmill test.
  Patients will have to do 3 walking sessions per week for a total duration of 12 weeks.
Benefit of music therapy (delivered by the BeatMove device) in a three-month outpatient walking rehabilitation: Sham group. | Week 12
  Maximum walking distance defined as the walking distance to the point of maximum muscular pain requiring stopping, during a treadmill test.
  Patients will have to do 3 walking sessions per week for a total duration of 12 weeks.

SECONDARY OUTCOMES:
Systolic pressure index at the toe at rest. Experimental group | Day 0 at the time of consultation
  Evaluation of the impact of music therapy on distal perfusion via Systolic Pressure Index at the toe after 3 months of rehabilitation
Systolic pressure index at the toe at rest. Experimental group | Week 12
  Evaluation of the impact of music therapy on distal perfusion via Systolic Pressure Index at the toe after 3 months of rehabilitation
Systolic pressure index at the toe after effort. Experimental group | Day 0 at the time of consultation
  Evaluation of the impact of music therapy on distal perfusion via Systolic Pressure Index at the toe after 3 months of rehabilitation
Systolic pressure index at the toe after effort. Experimental group | Week 12
  Evaluation of the impact of music therapy on distal perfusion via Systolic Pressure Index at the toe after 3 months of rehabilitation
Systolic pressure index at the toe at rest. Sham group | Day 0 at the time of consultation
  Evaluation of the impact of music therapy on distal perfusion via Systolic Pressure Index at the toe after 3 months of rehabilitation
Systolic pressure index at the toe at rest. Sham group | Week 12
  Evaluation of the impact of music therapy on distal perfusion via Systolic Pressure Index at the toe after 3 months of rehabilitation
Systolic pressure index at the toe after effort. Sham group | Day 0 at the time of consultation
  Evaluation of the impact of music therapy on distal perfusion via Systolic Pressure Index at the toe after 3 months of rehabilitation
Systolic pressure index at the toe after effort. Sham group | Week 12
  Evaluation of the impact of music therapy on distal perfusion via Systolic Pressure Index at the toe after 3 months of rehabilitation
Results of the EQ-5D-5L questionnaire in the experimental group | Day 0 at the time of consultation
  Patients will complete the EQ-5D-5L quality of life questionnaire before starting the walking training program and after completing it.
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Results of the EQ-5D-5L questionnaire in the experimental group | Week 12
  Patients will complete the EQ-5D-5L quality of life questionnaire before starting the walking training program and after completing it.
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Results of the EQ-5D-5L questionnaire in the sham group | Day 0 at the time of consultation
  Patients will complete the EQ-5D-5L quality of life questionnaire before starting the walking training program and after completing it.
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Results of the EQ-5D-5L questionnaire in the sham group | Week 12
  Patients will complete the EQ-5D-5L quality of life questionnaire before starting the walking training program and after completing it.
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Phone call follow-up in the experimental group | Week 4
  Patients in both groups will be followed up by a telephone call, 1 call per month, to assess compliance with the training program and monitor proper use of the device.
  The following information will be be recorded during follow-up phone calls and will include any problems encountered with :
  * Using the smartphone,
  * Use of BeatMove
  * Use of ankle sensors
  * Physical problems encountered during rehabilitation sessions
  * Medical problems
  * The problem of time and organization
  * Motivation problem
  * Other problems
Phone call follow-up in the sham group | Week 4
  Patients in both groups will be followed up by a telephone call, 1 call per month, to assess compliance with the training program and monitor proper use of the device.
  The following information will be be recorded during follow-up phone calls and will include any problems encountered with :
  * Using the smartphone,
  * Use of BeatMove
  * Use of ankle sensors
  * Physical problems encountered during rehabilitation sessions
  * Medical problems
  * The problem of time and organization
  * Motivation problem
  * Other problems
Phone call follow-up in the experimental group | Week 8
  Patients in both groups will be followed up by a telephone call, 1 call per month, to assess compliance with the training program and monitor proper use of the device.
  The following information will be be recorded during follow-up phone calls and will include any problems encountered with :
  * Using the smartphone,
  * Use of BeatMove
  * Use of ankle sensors
  * Physical problems encountered during rehabilitation sessions
  * Medical problems
  * The problem of time and organization
  * Motivation problem
  * Other problems
Phone call follow-up in the sham group | Week 8
  Patients in both groups will be followed up by a telephone call, 1 call per month, to assess compliance with the training program and monitor proper use of the device.
  The following information will be be recorded during follow-up phone calls and will include any problems encountered with :
  * Using the smartphone,
  * Use of BeatMove
  * Use of ankle sensors
  * Physical problems encountered during rehabilitation sessions
  * Medical problems
  * The problem of time and organization
  * Motivation problem
  * Other problems
Phone call follow-up in the experimental group | Week 12
  Patients in both groups will be followed up by a telephone call, 1 call per month, to assess compliance with the training program and monitor proper use of the device.
  The following information will be be recorded during follow-up phone calls and will include any problems encountered with :
  * Using the smartphone,
  * Use of BeatMove
  * Use of ankle sensors
  * Physical problems encountered during rehabilitation sessions
  * Medical problems
  * The problem of time and organization
  * Motivation problem
  * Other problems
Phone call follow-up in the sham group | Week 12
  Patients in both groups will be followed up by a telephone call, 1 call per month, to assess compliance with the training program and monitor proper use of the device.
  The following information will be be recorded during follow-up phone calls and will include any problems encountered with :
  * Using the smartphone,
  * Use of BeatMove
  * Use of ankle sensors
  * Physical problems encountered during rehabilitation sessions
  * Medical problems
  * The problem of time and organization
  * Motivation problem
  * Other problems
Patient's logbook: Pre- and post-workout pain rating in the experimental group | Three sessions per week for 3 months throughout the training program
  The patient's appreciation of pre- and post-workout pain will be recorded on a Lickert scale from 0 to 10 in which 0 = no pain, 10 = unbearable pain.
Patient's logbook: Pre- and post-workout pain rating in the sham group | Three sessions per week for 3 months throughout the training program
  The patient's appreciation of pre- and post-workout pain will be recorded on a Lickert scale from 0 to 10 in which 0 = no pain, 10 = unbearable pain.
Patient's logbook: Pre- and post-workout evaluation of fatigue in the experimental group | Three sessions per week for 3 months throughout the training program
  Evaluation of fatigue before and after training (Lickert scale from 0 to 10 in which 0 = no fatigue, 10 = greatest possible fatigue).
Patient's logbook: Pre- and post-workout evaluation of fatigue in the sham group | Three sessions per week for 3 months throughout the training program
  Evaluation of fatigue before and after training (Lickert scale from 0 to 10 in which 0 = no fatigue, 10 = greatest possible fatigue).
Patient's logbook: Pre- and post-workout evaluation of motivation in the experimental group | Three sessions per week for 3 months throughout the training program
  Evaluation of motivation before and after training (Lickert scale from 0 to 10 in which 0 = no motivation, 10 = greatest possible motivation).
Patient's logbook: Pre- and post-workout evaluation of motivation in the sham group | Three sessions per week for 3 months throughout the training program
  Evaluation of motivation before and after training (Lickert scale from 0 to 10 in which 0 = no motivation, 10 = greatest possible motivation).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, France